CLINICAL TRIAL: NCT01112917
Title: VenaTech Convertible Vena Cava Filter U.S. Multi-Center Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: B. Braun Interventional Systems, Inc (Industry)
Collaborators: Bright Research Partners (Industry); NAMSA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CL-104
Record Dates: First submitted 2010-04-08; First posted 2010-04-29 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-06

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VenaTech Convertible Vena Cava Filter (Experimental): Implantation of the VenaTech Convertible Filter. The filter is pre-loaded in a cartridge (syringe) and provided as a system with introducer accessories and instructions to accommodate delivery and implantation either using the femoral or jugular approach.
  Interventions: Device: VenaTech Convertible Vena Cava Filter; Procedure: Vena Cava Filter Conversion

INTERVENTIONS:
Device: VenaTech Convertible Vena Cava Filter — Prevention of Pulmonary Embolism
Procedure: Vena Cava Filter Conversion — Conversion of VenaTech Convertible filter to open configuration.

SUMMARY:
The investigation is designed to verify that clinical use of the vena cava filter does not raise new questions of safety or effectiveness compared to currently-marketed permanent filters.

DETAILED DESCRIPTION:
The investigation was designed as a multi-center, prospective, single-arm, historical (literature) controlled clinical study of VenaTech Convertible filter safety and performance in 75 subjects in whom the filter has been implanted, converted, and followed for 6-months. The study could enroll up to 323 patients to ensure 75 converted subjects with 6 months of follow-up data. Converted subjects were followed at 30-days, 3-months, and 6-months post conversion. Subjects that were unable to undergo conversion were followed at 6-months post filter implant (permanent filtration subjects).

Study subjects were to be identified from the pool of candidates with a time-limited risk for pulmonary embolism. Subjects who signed the informed consent were evaluated to determine eligibility for the study based on the inclusion and exclusion criteria. Following completion of baseline procedures including a bilateral Doppler ultrasound of the legs to assess for baseline DVT and contrast venacavography to assess baseline IVC diameter, subjects underwent implantation of the VenaTech Convertible filter.

After device implant, a clinical assessment was completed to determine eligibility for filter conversion. This assessment was done at an interval post-implant and frequency per the investigator's discretion, often with input from the primary care physician. If the clinician determined the subject was no longer at risk for pulmonary embolism, there was no thrombus in or below the filter, and there was no clinically significant deep vein thrombosis (DVT) in the legs, the filter could be converted. After conversion, subjects were followed at 30 days and 3-months by telephone, and at a 6-months post-conversion office visit with imaging (KUB or spot film and Doppler or CT).

If during the conversion clinical assessment(s), the subject remained at risk for pulmonary embolism, additional conversion assessment(s) were completed per the investigator's discretion until the filter was either converted or the subject was determined to require permanent filtration.

At 6-months post-implant, if a study subject's filter had not been converted, no further conversion assessments were to be performed and no attempts were to be made to convert the filter as part of the study. The 6-month post filter implant visit was the final follow-up for nonconverted subjects, which also included imaging (KUB or spot film and Doppler or CT). The study protocol allowed the investigators flexibility as to the best IVC imaging modality based on the condition and anatomy of the subject.

The core laboratory reviewed all screening/baseline, filter implantation, conversion eligibility assessment, conversion, and 6-month follow-up images, with the exception of the ultrasounds. (The core laboratory recommended ultrasound images be evaluated by the expert sonographers at the sites). Additionally, any images taken as a result of a suspected filter-related adverse event or technical complication, with the exception of ultrasounds, were also sent to the core laboratory for review.

ELIGIBILITY:
Inclusion Criteria:

* The subject is 18 years of age or older
* The subject is at a time-limited risk of pulmonary embolism as judged by the implanting or referring physician
* In the physician's judgment, the subject requires prevention of pulmonary embolism and placement of a vena cava filter is indicated because anticoagulants are contraindicated, or the subject has experienced failure of anticoagulant therapy in thromboembolic diseases in the past, or the subject requires emergency treatment following massive pulmonary embolism where anticipated benefits of conventional therapy are reduced
* The subject, or their legal representative, is willing and able to provide informed consent
* The subject is willing and able to comply with the requirements of the study protocol, including the predefined follow-up visit evaluations
* The subject's vena cava diameter is ≤ 28 mm as evaluated by contrast venacavography and corrected for magnification

Exclusion Criteria:

* The subject is a female of childbearing potential and known to be, or suspected to be, pregnant (verified with a urine/blood pregnancy test), or unwilling to use an acceptable form of birth control for as long as the device is implanted
* The subject is severely disabled and his/her life expectancy appears limited according to the investigator's opinion (≤ 6 months)
* The subject already has an implanted vena cava filter
* The subject has contrast allergy to both iodinated contrast and non-iodinated contrast materials
* The subject has a duplicated IVC
* The subject is bacteremic
* The subject has an active malignancy with associated hypercoagulability or mortality likely preventing the VenaTech Convertible filter from being converted within 6 months of implant
* The subject would be unavailable for follow-up
* Filter implantation using the right internal jugular or femoral veins is not possible
* There is no location available in the infrarenal inferior vena cava for placement of the VenaTech Convertible vena cava filter (assessed using contrast venacavography)
* The subject is currently participating in another clinical study or has participated in one within the last 30 days or plans to participate in one during the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2011-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William S Rilling, MD, Principal Investigator — Froedtert Hospital
Locations (11):
- United States (11):
  - Baptist Hospital of Miami, Miami, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Adventist Health System, Hinsdale, Illinois
  - Beaumont Health System, Royal Oak, Michigan
  - North Shore University Hospital - Manhasset, Manhasset, New York
  - Weill Cornell Medical College - New York Presbyterian Hospital, New York, New York
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Virginia Health Systems, Charlottesville, Virginia
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vena Caval Filter Consensus Conference. Recommended reporting standards for vena caval filter placement and patient follow-up. J Vasc Surg. 1999 Sep;30(3):573-9. No abstract available. PMID 10477662
- [Background] Grassi CJ, Swan TL, Cardella JF, Meranze SG, Oglevie SB, Omary RA, Roberts AC, Sacks D, Silverstein MI, Towbin RB, Lewis CA; Society of Interventional Radiology Standards of Practice Committee. Quality improvement guidelines for percutaneous permanent inferior vena cava filter placement for the prevention of pulmonary embolism. J Vasc Interv Radiol. 2003 Sep;14(9 Pt 2):S271-5. No abstract available. PMID 14514832

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants were first implanted with the VenaTech Convertible Filter. After the implantation, the study investigators assessed whether participants were eligible for conversion of the filter or required permanent filtration. If a subject was not eligible for conversion at 6-months, they were considered a permanent filtration subject.
Groups:
- VenaTech Convertible Filter - Converted Filter: VenaTech Convertible Vena Cava Filter: Prevention of Pulmonary Embolism
  Vena Cava Filter Conversion: Conversion of VenaTech Convertible filter to open configuration.
- VenaTech Convertible Filter - Permanent Filtration: VenaTech Convertible Vena Cava Filter: Prevention of Pulmonary Embolism
Period: Overall Study
Arm/Group | VenaTech Convertible Filter - Converted Filter | VenaTech Convertible Filter - Permanent Filtration
Started | 96 | 53
Completed | 89 | 38
Not Completed | 7 | 15
Not completed — Death | 2 | 11
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Unable to Convert Filter | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- VenaTech Convertible Filter: VenaTech Convertible Vena Cava Filter: Prevention of Pulmonary Embolism
  Vena Cava Filter Conversion: Conversion of VenaTech Convertible filter to open configuration.
Arm/Group | VenaTech Convertible Filter
Number analyzed (Participants) | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 145
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 125
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 149

OUTCOME MEASURES:

1. Primary Outcome: Technical Success
Description: Technical success is defined as filter conversion without the loss of filter head components in the vasculature or incomplete opening of filtering legs. Further, in the analysis of the data, the sponsor did not count any filters as a 'technically' successful conversion when the operator was unable to snare the filter hook during an attempted conversion.
Time Frame: 6-months
Measure: Number; unit: participants
Groups:
- VenaTech Convertible Filter - Converted Filters: VenaTech Convertible Vena Cava Filter: Prevention of Pulmonary Embolism
  Vena Cava Filter Conversion: Conversion of VenaTech Convertible filter to open configuration.
Arm/Group | VenaTech Convertible Filter - Converted Filters
Number analyzed (Participants) | 96
participants | 89

2. Secondary Outcome: Major Device-Related Adverse Events in Converted Subjects
Time Frame: 6-months
Population: There was one subject (007-006) excluded as no 6-month images were available although a 6-month assessment was conducted.
Measure: Number; unit: participants
Arm/Group | VenaTech Convertible Filter - Converted Filters
Number analyzed (Participants) | 88
participants | 0

ADVERSE EVENTS:
Time Frame: 6-Month Follow-up Period (through 6-months post-implant or post-filter conversion)
Description: The "Other" adverse events were not broken down into separate specific Adverse Events, so are presented all under the "Other" category.
Arm/Group | VenaTech Convertible Filter
Serious Adverse Events (participants affected / at risk) | 63/149
Other Adverse Events (participants affected / at risk) | 77/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VenaTech Convertible Filter (N=149)
Caval Thrombosis or Caval Occlusion (Blood and lymphatic system disorders) | 4 (4)
Compromise of Cardiac Valve Function due to Filter Embolization (Blood and lymphatic system disorders) | 1 (1)
Death (General disorders) | 13 (13)
Deep Vein Thrombosis (DVT) (Blood and lymphatic system disorders) | 4 (8)
Infection, including access site infection (Infections and infestations) | 3 (3)
Pulmonary embolism (Blood and lymphatic system disorders) | 1 (1)
Other (General disorders) | 57 (89)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VenaTech Convertible Filter (N=149)
Access site thrombosis (Blood and lymphatic system disorders) | 1 (1)
Caval Thrombosis or Caval Occlusion (Blood and lymphatic system disorders) | 1 (1)
Deep Vein Thrombosis (DVT) (Blood and lymphatic system disorders) | 11 (15)
Infection, including access site infection (Infections and infestations) | 1 (1)
Other (General disorders) | 70 (166)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days